CLINICAL TRIAL: NCT00078949
Title: Phase III Study Of Gemcitabine, Dexamethasone, And Cisplatin Compared To Dexamethasone, Cytarabine, And Cisplatin Plus/Minus Rituximab [(R)-GDP vs (R)-DHAP] As Salvage Chemotherapy For Patients With Relapsed Or Refractory Aggressive Histology Non-Hodgkin's Lymphoma Prior To Autologous Stem Cell Transplant And Followed By Maintenance Rituximab vs Observation
Brief Title: Chemotherapy Before Autologous Stem Cell Transplantation +/- Rituximab in Relapsed or Refractory Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY12; CAN-NCIC-LY12; CDR0000353203 (Other: PDQ); NCT00089817 (obsolete NCT alias)
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2020-03

CONDITIONS: Lymphoma
Keywords: anaplastic large cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; angioimmunoblastic T-cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Immunoblastic Lymphadenopathy | interventions — Rituximab; Cisplatin; Cytarabine; Dexamethasone; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Salvage arm I (Experimental): Patients receive cisplatin IV over 60 minutes on day 1, dexamethasone IV or orally on days 1-4, and gemcitabine IV over 30 minutes on days 1 and 8.
  Interventions: Drug: cisplatin; Drug: dexamethasone; Drug: gemcitabine hydrochloride
- Salvage arm II (Experimental): Patients receive cisplatin IV over 24 hours on day 1, dexamethasone as in arm I, and cytarabine IV over 3 hours every 12 hours for a total of 2 doses on day 2.
  Interventions: Drug: cisplatin; Drug: cytarabine; Drug: dexamethasone
- Maintenance arm I (Experimental): Beginning on day 28 posttransplantation, patients receive rituximab IV once every 2 months for 6 doses (a total of 12 months) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab
- Maintenance arm II (No Intervention): Patients undergo observation only.

INTERVENTIONS:
Biological: rituximab — Given IV
  Arms: Maintenance arm I
Drug: cisplatin — Given IV
  Arms: Salvage arm I; Salvage arm II
Drug: cytarabine — Given IV
  Arms: Salvage arm II
Drug: dexamethasone — Given IV
  Arms: Salvage arm I; Salvage arm II
Drug: gemcitabine hydrochloride — Given IV
  Arms: Salvage arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as dexamethasone, cisplatin, gemcitabine, and cytarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with autologous stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Giving rituximab as maintenance therapy after stem cell transplantation may kill any remaining cancer cells. It is not yet known which salvage chemotherapy regimen is more effective before autologous stem cell transplantation in treating relapsed or refractory non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying salvage chemotherapy using dexamethasone, cisplatin, and gemcitabine to see how well it works compared to dexamethasone, cisplatin, and cytarabine given before autologous stem cell transplantation in treating patients with relapsed or refractory aggressive non-Hodgkin's lymphoma. This trial also is studying giving rituximab as maintenance therapy to see how well it works compared to no further therapy after stem cell transplantation. Rituximab was added to both salvage treatment arms for CD20+ patients in a protocol amendment in 2005.

DETAILED DESCRIPTION:
OBJECTIVES:

Salvage therapy

Primary

* Compare the response rate and transplantation rate in patients with relapsed or refractory aggressive non-Hodgkin's lymphoma when treated with salvage chemotherapy comprising dexamethasone, cisplatin, and gemcitabine with or without rituximab vs a standard platinum-based regimen (dexamethasone, cisplatin, and high-dose cytarabine with or without rituximab).
* To compare the transplantation rates of the two protocol salvage regimens.

Secondary

* Compare the event-free and overall survival of patients treated with these regimens.
* Compare the success rate of these regimens, in terms of getting patients to autologous stem cell transplantation and successful mobilization after high-dose chemotherapy.
* Compare the quality of life of patients treated with these salvage regimens.
* Compare the toxic effects of these salvage regimens in these patients.
* Compare resource utilization for patients treated with these salvage regimens.
* Compare relative medical and societal costs of these salvage regimens with outcomes in these patients.

Maintenance therapy

Primary

* Compare the 2-year event-free survival of patients with CD20+ B-cell lymphoma treated with maintenance rituximab after these salvage regimens and autologous stem cell transplantation to those patients who received no further treatment.

Secondary

* Compare the 2-year survival of patients treated with or without maintenance rituximab.
* Compare the toxic effects of rituximab vs observation alone in these patients.

OUTLINE: This is a randomized, multicenter study. For salvage therapy, patients are stratified according to participating center, International Prognostic Index score at relapse/study entry (0 or 1 vs 2 vs ≥ 3), immunophenotype (B cell vs T cell), response to or response duration after initial chemotherapy (no response or progressive disease vs > 1 year vs ≤ 1 year), and prior rituximab (yes vs no). For maintenance therapy, patients are stratified according to participating center, salvage therapy treatment randomization (with or without rituximab, cisplatin, dexamethasone, and gemcitabine vs with or without rituximab, cisplatin, dexamethasone, and cytarabine), response to salvage therapy (complete response [CR] and CR unconfirmed [CRu] vs partial response [PR] vs stable disease [SD]), and prior rituximab (yes vs no).

* Salvage therapy: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive cisplatin IV over 60 minutes on day 1, dexamethasone IV or orally on days 1-4, and gemcitabine IV over 30 minutes on days 1 and 8. Patients with CD20+ B cell lymphoma receive rituximab IV over 1.5-6 hours on day 1.
  * Arm II: Patients receive cisplatin IV over 24 hours on day 1, dexamethasone as in arm I, and cytarabine IV over 3 hours every 12 hours for a total of 2 doses on day 2. Patients with CD20+ B cell lymphoma receive rituximab IV over 1.5-6 hours on day 1.

In both arms, treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are reassessed after 2 courses. Patients with progressive disease are removed from study. Patients with a CR, CRu, or PR proceed to autologous stem cell transplantation (ASCT). Patients with SD may proceed to ASCT or receive 1 additional course of salvage therapy at the discretion of the investigator. Patients receiving an additional course of salvage therapy are then reassessed after the completion of therapy. Patients with progressive disease are removed from study. Patients with a PR proceed to ASCT. Patients with SD may proceed to ASCT or be followed off study at the discretion of the investigator.

* ASCT: Responding patients (or those with stable disease, if that is the center's policy)undergo mobilization, stem cell harvest, and subsequent ASCT. Patients with CD20+ B-cell disease are randomized to maintenance therapy or observation.
* Maintenance therapy: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Beginning on day 28 posttransplantation, patients receive rituximab IV once every 2 months for 6 doses (a total of 12 months) in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients undergo observation only. Quality of life is assessed at baseline, days 1 and 10 of course 2, day 1 of course 3 (if given), on the last day of salvage therapy (or the first day of mobilization, if given), and at 1 month posttransplantation.

Patients who undergo ASCT are followed at months 1, 3, 7, 13, 19, and 25 and then annually thereafter. Patients who complete salvage therapy, but do not undergo ASCT are followed at months 4, 8, 14, 20, and 26 and then annually thereafter. Patients who relapse or progress are followed every 6 months until 25 months from ASCT or 26 months from completion of salvage therapy and then annually thereafter.

PROJECTED ACCRUAL: A total of 637 patients will be accrued for this study within 3-4 years for the first randomization, and 240 transplanted CD20+ patients will be needed for the second randomization.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive non-Hodgkin's lymphoma of 1 of the following subtypes:

  * Diffuse large cell lymphoma (includes primary mediastinal B-cell lymphoma and T-cell-rich B-cell lymphoma)
  * Prior indolent lymphoma (e.g., follicular center cell lymphoma; marginal zone lymphoma, including extranodal mucosa-associated lymphoid tissue [MALT] lymphoma; and lymphoplasmacytoid lymphoma) with transformation to diffuse large B-cell lymphoma at relapse

    * Must be histologically confirmed
    * No transformed lymphoma at diagnosis with subsequent indolent histology without transformation at relapse
  * Peripheral T-cell lymphoma
  * Anaplastic large cell lymphoma
  * Small noncleaved Burkitt-like lymphoma
* T-cell or B-cell lineage confirmed by immunohistochemistry
* Clinically or radiologically documented disease meeting either of the following criteria:

  * Measurable disease, defined as at least 1 bidimensionally measurable site of disease using clinical exam, CT scan, or MRI

    * Lymph nodes must be > 1.5 cm by physical exam or CT scan
    * Other non-nodal lesions must be ≥ 1.0 cm by physical exam, CT scan, or MRI
    * Bone lesions are not considered measurable
  * Evaluable disease, defined as only nonmeasurable disease, including any of the following:

    * Marrow infiltration
    * Cytology-confirmed ascites or effusions
    * Bony involvement
    * Enlarged liver or spleen
    * Unidimensionally measurable intrathoracic or abdominal masses
* Previously treated with 1, and only 1, chemotherapy regimen including an anthracycline and excluding cisplatin, cytarabine, and gemcitabine
* No uncontrolled CNS involvement by lymphoma

  * No CNS disease at time of relapse
  * CNS disease diagnosed at initial presentation allowed provided a complete response for CNS disease was achieved and maintained

PATIENT CHARACTERISTICS:

Age

* 16 to 65

Performance status

* ECOG 0-3

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT ≤ 2.5 times ULN (5 times ULN if liver involvement with lymphoma)
* Hepatitis B status known (for patients with a history of hepatitis B or who are at high risk of hepatitis B infection)

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No significant cardiac dysfunction or cardiovascular disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to complete quality of life questionnaires
* HIV negative
* No active, uncontrolled bacterial, fungal, or viral infection
* No other malignancy within the past 5 years except adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* No other concurrent serious illness or medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Chemotherapy
* Prior rituximab allowed

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior IV chemotherapy
* No prior high-dose chemotherapy with stem cell transplantation

Endocrine therapy

* No concurrent corticosteroids except for physiologic replacement

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered

  * Exceptions may be made for low-dose, non-myelosuppressive radiotherapy
* No prior radiotherapy to more than 25% of functioning bone marrow
* Involved-field radiotherapy may be given to areas of bulky disease at relapse (≥ 5 cm) after stem cell transplantation, according to the center's policy

Surgery

* At least 2 weeks since prior major surgery

Other

* No other concurrent anticancer therapy
* No other concurrent experimental agents

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 849 (Actual)
Dates: Start 2003-08-27 (Actual); Primary Completion 2013-07-29 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Crump, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada; Massimo Federico, MD, Study Chair — Azienda Ospedaliero-Universitaria di Modena
Locations (27):
- United States (5):
  - Rush-Presbyterian-St. Luke's Medical Centre, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Cincinnati, Barrett Cancer Centre, Cincinnati, Ohio
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
- The Queen Elizabeth Hospital, Woodville, South Australia, Australia
- Canada (21):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta A, Hay AE, Crump M, Djurfeldt MS, Zhu L, Cheung MC, Shepherd LE, Chen BE, Booth CM. Contact Days Associated With Cancer Treatments in the CCTG LY.12 Trial. Oncologist. 2023 Sep 7;28(9):799-803. doi: 10.1093/oncolo/oyad128. PMID 37226534
- [Result] Crump M, Kuruvilla J, Couban S, MacDonald DA, Kukreti V, Kouroukis CT, Rubinger M, Buckstein R, Imrie KR, Federico M, Di Renzo N, Howson-Jan K, Baetz T, Kaizer L, Voralia M, Olney HJ, Turner AR, Sussman J, Hay AE, Djurfeldt MS, Meyer RM, Chen BE, Shepherd LE. Randomized comparison of gemcitabine, dexamethasone, and cisplatin versus dexamethasone, cytarabine, and cisplatin chemotherapy before autologous stem-cell transplantation for relapsed and refractory aggressive lymphomas: NCIC-CTG LY.12. J Clin Oncol. 2014 Nov 1;32(31):3490-6. doi: 10.1200/JCO.2013.53.9593. Epub 2014 Sep 29. PMID 25267740
- [Derived] Gupta A, Thomas T, Hay AE, Crump M, Djurfeldt MS, Cheung MC, Prica A, Shepherd LE, Chen BE, Booth CM. The association of health care contact days with economic measures in the CCTG LY.12 trial. Oncologist. 2025 Jun 4;30(6):oyaf165. doi: 10.1093/oncolo/oyaf165. PMID 40503814
- [Derived] Assouline S, Li S, Gisselbrecht C, Fogarty P, Hay A, van den Neste E, Shepherd LE, Schmitz N, Baetz T, Keating A, Robinson S, Seftel M, Stelitano C, Djurfeldt MS, Meyer R, Chen BE, Crump M. The conditional survival analysis of relapsed DLBCL after autologous transplant: a subgroup analysis of LY.12 and CORAL. Blood Adv. 2020 May 12;4(9):2011-2017. doi: 10.1182/bloodadvances.2020001646. PMID 32396614
- [Derived] Bosch M, Akhter A, Chen BE, Mansoor A, Lebrun D, Good D, Crump M, Shepherd L, Scott DW, Stewart DA. A bioclinical prognostic model using MYC and BCL2 predicts outcome in relapsed/refractory diffuse large B-cell lymphoma. Haematologica. 2018 Feb;103(2):288-296. doi: 10.3324/haematol.2017.179309. Epub 2017 Nov 2. PMID 29097500
- [Derived] Davison K, Chen BE, Kukreti V, Couban S, Benger A, Berinstein NL, Kaizer L, Desjardins P, Mangel J, Zhu L, Djurfeldt MS, Hay AE, Shepherd LE, Crump M. Treatment outcomes for older patients with relapsed/refractory aggressive lymphoma receiving salvage chemotherapy and autologous stem cell transplantation are similar to younger patients: a subgroup analysis from the phase III CCTG LY.12 trial. Ann Oncol. 2017 Mar 1;28(3):622-627. doi: 10.1093/annonc/mdw653. PMID 27993811
- [Derived] Kuruvilla J, MacDonald DA, Kouroukis CT, Cheung M, Olney HJ, Turner AR, Anglin P, Seftel M, Ismail WS, Luminari S, Couban S, Baetz T, Meyer RM, Hay AE, Shepherd L, Djurfeldt MS, Alamoudi S, Chen BE, Crump M. Salvage chemotherapy and autologous stem cell transplantation for transformed indolent lymphoma: a subset analysis of NCIC CTG LY12. Blood. 2015 Aug 6;126(6):733-8. doi: 10.1182/blood-2015-01-622084. Epub 2015 Jun 24. PMID 26109202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 619 patients in the first randomization. Only a selected subset of patient (N = 230) were randomized in period 2 of this study. Total sample size N = 849
Groups:
- Salvage GDP: Patients receive cisplatin IV over 60 minutes on day 1, dexamethasone IV or orally on days 1-4, and gemcitabine IV over 30 minutes on days 1 and 8.
  cisplatin: Given IV
  dexamethasone: Given IV
  gemcitabine hydrochloride: Given IV
- Salvage DHAP: Patients receive cisplatin IV over 24 hours on day 1, dexamethasone as in arm I, and cytarabine IV over 3 hours every 12 hours for a total of 2 doses on day 2.
  cisplatin: Given IV
  cytarabine: Given IV
  dexamethasone: Given IV
- Maintenance: Beginning on day 28 posttransplantation, patients receive rituximab IV once every 2 months for 6 doses (a total of 12 months) in the absence of disease progression or unacceptable toxicity.
  rituximab: Given IV
- Observation: Patients undergo observation only.
Period: Overall Study
Arm/Group | Salvage GDP | Salvage DHAP | Maintenance | Observation
Started | 310 | 309 | 115 | 115
Completed | 306 | 304 | 112 | 112
Not Completed | 4 | 5 | 3 | 3
Not completed — No treated | 4 | 5 | 3 | 3

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Salvage GDP | Salvage DHAP | Maintenance | Observation | Total
Number analyzed (Participants) | 310 | 309 | 115 | 115 | 849
Age, Continuous [Median (Full Range); unit: years] | 55 [19 to 71] | 55 [23 to 74] | 54 [25 to 68] | 55 [30 to 69] | 55 [19 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 118 | 44 | 48 | 332
  Male | 188 | 191 | 71 | 67 | 517

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Patients After 2 Courses of Chemotherapy
Description: The overall response rate by arm is calculated as total number of responders (CR + CRu + PR) / (all patients in the ITT analysis population).
Time Frame: After 2 cycle of treatment
Population: ITT population
Measure: Number; unit: percentage of response
Arm/Group | Salvage GDP | Salvage DHAP
Number analyzed (Participants) | 310 | 309
percentage of response | 45.2 | 44.0
Statistical Analysis 1: Comparison: Salvage GDP vs Salvage DHAP; Test type: Non-Inferiority or Equivalence — The literature has suggested that the ORR is approximately 50% for this patient population treated with DHAP. The treatment difference is defined as the response rate for the DHAP arm minus that of GDP arm. We would consider GDP to be non-inferior to DHAP if we are 95% sure that the true difference is less than 10%. In order to rule out that the 10% difference with 80% power, we need to accrue a total of 630 eligible patients. The actual sample size for this final analysis is 619 patients; p = 0.005, Cochran-Mantel-Haenszel — p-value for non-inferiority; Risk Difference (RD) = -1.2, 95% CI 2-sided [-9.0 to 6.7]

2. Primary Outcome: Transplantation Rate of Patients After 2 Courses of Chemotherapy
Description: Transplantation rate is defined as the number of patients who respond sufficiently to protocol salvage chemotherapy to be planned for transplantation minus those who do not meet the endpoint of successful transplantation, divided by the number of all randomized patients
Time Frame: During period 1 (salvage chemotherapy)
Measure: Number; unit: percentage of transplantation
Arm/Group | Salvage GDP | Salvage DHAP
Number analyzed (Participants) | 310 | 309
percentage of transplantation | 51.0 | 48.9
Statistical Analysis 1: Comparison: Salvage GDP vs Salvage DHAP; Test type: Superiority or Other; p = 0.55, Cochran-Mantel-Haenszel; Risk Difference (RD) = -2.1, 95% CI [-10.0 to 5.8]

3. Primary Outcome: Event-free Survival of Patients on Maintenance Randomization (Period 2)
Description: Number of patients who develop EFS event during maintenance randomization (period 2)
Time Frame: during the period 2 (up to10 years)
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Maintenance | Observation
Number analyzed (Participants) | 115 | 115
participants | 53 | 65
Statistical Analysis 1: Comparison: Maintenance vs Observation; It was estimated that 240 patients will be eligible for the maintenance question, and randomized with a 1:1 ratio to either rituximab or observation. It is expected that the 2-year event-free survival will be 50% on the observation arm. In order to detect a 15% difference in the 2-year event-free survival with an 80% power using a two-sided 5% level test, 142 events are required to detect an HR of 0.622; Test type: Superiority or Other; p = 0.17, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.52 to 1.12]

4. Secondary Outcome: Toxic Effect
Description: Number of patients affected by adverse events graded according to CTC Version 2.0. See adverse event (others) for details.
Time Frame: 48 months
Population: All patients who received the protocol treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Salvage GDP | Salvage DHAP | Maintenance | Observation
Number analyzed (Participants) | 306 | 304 | 112 | 112
Participants | 36 | 26 | 16 | 8

ADVERSE EVENTS:
Time Frame: 8.5 year
Description: Serious and Other Adverse Events were assessed in participants who received protocol treatment. All-cause mortality was collected for all enrolled participants
Arm/Group | Salvage GDP | Salvage DHAP | Maintenance | Observation
All-Cause Mortality (participants affected / at risk) | 177/310 | 181/309 | 39/115 | 42/115
Serious Adverse Events (participants affected / at risk) | 36/306 | 26/304 | 16/112 | 8/112
Other Adverse Events (participants affected / at risk) | 287/306 | 293/304 | 98/112 | 90/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Salvage GDP (N=306) | Salvage DHAP (N=304) | Maintenance (N=112) | Observation (N=112)
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
DIC (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 11 | 3 | 1
Edema (Cardiac disorders) | 1 | 0 | 0 | 0
Ischemia/infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 2 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2 | 0
Melena/GI bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal bleeding (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Hematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0
Pain-Other (General disorders) | 2 | 0 | 1 | 1
Other (Immune system disorders) | 1 | 1 | 0 | 0
Other (Immune system disorders) | 3 | 0 | 0 | 1
Fever (Immune system disorders) | 3 | 3 | 2 | 0
Other (Immune system disorders) | 1 | 0 | 1 | 0
Other (Immune system disorders) | 1 | 0 | 0 | 0
Wound-infectious (Infections and infestations) | 1 | 0 | 0 | 0
Granulocytes (Investigations) | 2 | 0 | 1 | 0
Lymphopenia (Investigations) | 1 | 0 | 0 | 0
Platelets (Investigations) | 0 | 1 | 0 | 0
Leukocytes (total WBC) (Investigations) | 1 | 1 | 0 | 0
Cardiac troponin T (Investigations) | 0 | 1 | 0 | 0
Creatinine (Investigations) | 1 | 2 | 1 | 0
SGPT (ALT) (Investigations) | 1 | 0 | 0 | 0
SGOT (AST) (Investigations) | 1 | 0 | 0 | 0
Bilirubin (Investigations) | 1 | 0 | 0 | 0
Weight loss (Investigations) | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 3 | 3
Hemorrhage/bleeding (Nervous system disorders) | 1 | 0 | 0 | 0
Speech impairment (Nervous system disorders) | 2 | 0 | 0 | 0
Neuropathy-sensory (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 1 | 0
Thrombosis/embolism (Vascular disorders) | 5 | 2 | 3 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Salvage GDP (N=306) | Salvage DHAP (N=304) | Maintenance (N=112) | Observation (N=112)
Febrile neutropenia (Blood and lymphatic system disorders) | 28 | 71 | 10 | 3
Edema (Cardiac disorders) | 39 | 64 | 8 | 9
Inner ear/hearing (Ear and labyrinth disorders) | 50 | 76 | 14 | 12
Blurred vision (Eye disorders) | 21 | 15 | 5 | 3
Constipation (Gastrointestinal disorders) | 133 | 113 | 10 | 14
Diarrhea (Gastrointestinal disorders) | 64 | 85 | 19 | 11
Dysphagia (Gastrointestinal disorders) | 17 | 17 | 12 | 3
Dyspepsia/heartburn (Gastrointestinal disorders) | 59 | 51 | 17 | 10
Nausea (Gastrointestinal disorders) | 172 | 221 | 22 | 14
Stomatitis (Gastrointestinal disorders) | 61 | 70 | 7 | 2
Vomiting (Gastrointestinal disorders) | 95 | 151 | 18 | 8
Other (Gastrointestinal disorders) | 4 | 6 | 8 | 0
Abdominal pain (Gastrointestinal disorders) | 65 | 47 | 22 | 14
Fatigue (General disorders) | 225 | 201 | 65 | 59
Rigors, chills (General disorders) | 10 | 21 | 6 | 5
Chest pain (General disorders) | 19 | 27 | 5 | 7
Pain-Other (General disorders) | 21 | 23 | 10 | 4
Fever (Immune system disorders) | 45 | 74 | 14 | 12
Infection w/o neutropen (Infections and infestations) | 64 | 58 | 50 | 39
Weight loss (Investigations) | 18 | 15 | 12 | 7
Anorexia (Metabolism and nutrition disorders) | 77 | 94 | 17 | 16
Dehydration (Metabolism and nutrition disorders) | 17 | 22 | 3 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 18 | 3 | 2
Muscle weakness (Musculoskeletal and connective tissue disorders) | 23 | 20 | 6 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 15 | 20 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 49 | 42 | 25 | 24
Bone pain (Musculoskeletal and connective tissue disorders) | 33 | 32 | 17 | 17
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 46 | 41 | 6 | 2
Taste disturbance (Nervous system disorders) | 28 | 43 | 10 | 11
Dizziness (Nervous system disorders) | 39 | 33 | 12 | 5
Neuropathy-motor (Nervous system disorders) | 30 | 13 | 5 | 3
Neuropathy-sensory (Nervous system disorders) | 106 | 74 | 25 | 28
Syncope (Nervous system disorders) | 7 | 16 | 0 | 1
Headache (Nervous system disorders) | 59 | 72 | 10 | 6
Neuropathic pain (Nervous system disorders) | 7 | 9 | 9 | 8
Anxiety (Psychiatric disorders) | 40 | 30 | 10 | 8
Insomnia (Psychiatric disorders) | 61 | 54 | 13 | 10
Depression (Psychiatric disorders) | 20 | 13 | 7 | 7
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 10 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 16 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 55 | 61 | 38 | 19
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 18 | 17 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 65 | 69 | 19 | 24
Sweating (Skin and subcutaneous tissue disorders) | 51 | 33 | 13 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 31 | 42 | 13 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 14 | 7 | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 61 | 38 | 10 | 15
Other (Skin and subcutaneous tissue disorders) | 7 | 6 | 6 | 4
Hypotension (Vascular disorders) | 14 | 25 | 4 | 1
Thrombosis/embolism (Vascular disorders) | 24 | 24 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No